CLINICAL TRIAL: NCT00570583
Title: Clinical Studies of Mental Illness Not Involving Treatment Development, Efficacy, or Effectiveness Trials Phenotype-genotype Predictors of Cognitive Outcomes in Geriatric Depression
Brief Title: Neurocognitive Outcomes of Depression in the Elderly
Acronym: NCODE
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00006424; 1R01MH108560-01 (NIH); 0625
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Major Depression; Dementia
Keywords: Depression; Cognitive impairment; Dementia; Neuroimaging; Genetics
MeSH Terms: conditions — Depressive Disorder, Major; Dementia; Depression; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Depressed: Older individuals with major depression
- Non-depressed: Older individuals without psychiatric disorder

SUMMARY:
Late-life depression (LLD) and cognitive impairment (CI) are significant public health problems among older adults, and their co-occurrence markedly increases disease burden and dementia risk. This highlights the importance of identifying and treating CI in LDD; however, current lack of reliable prognostic information from clinical, neuroimaging, and genetic data impedes research on targeted prevention and treatment. Two critical ways to close current knowledge gaps in predicting cognitive diagnostic outcomes of LLD involve: 1) increasing the number of diagnostic cases available to existing studies, and 2) using those studies to identify clinical, imaging, and genetic predictors that will improve future diagnosis. We intend to do both in the current proposal. We plan to study the following SPECIFIC AIMS:

Aim 1: Identify baseline clinical-behavioral predictors of cognitive diagnostic outcomes in LLD.

Working hypothesis: During acute LLD, CN will be associated with more frequent EOD and higher negative life stress than PCI and AD; PCI will be associated with EOD and higher frailty than CN and AD; AD will be associated with LOD, greater appetite loss, lower anxiety, and greater memory impairment than CN and PCI.

Aim 2: Use multimodal neuroimaging at baseline to identify patterns associated with cognitive diagnostic outcomes in individuals with LLD. Working Hypothesis: CN will be associated with greater white matter integrity compared with PCI and AD; PCI will be associated with lower white matter integrity and network abnormalities in anterior cingulate cortex compared with CN; AD will be associated with lower hippocampal volume compared with CN and PCI.

Aim 3: (exploratory): Explore interrelationships among candidate genes, cognitive diagnostic outcomes, and proposed phenotypic components relevant to LLD. Exploratory Hypotheses: 1) COMT val158met polymorphism will be associated with CN; 2) 5-HTTPRL and APOE ε2 polymorphisms will be associated with frailty; 3) genetic variation (SNPs) in TPH2 and AGTR1 will be associated with risk factors of AD: LOD, episodic memory, hippocampal volume, and appetite loss.

DETAILED DESCRIPTION:
Central hypothesis: the 5-year likelihood of each cognitive diagnostic outcome is associated with distinct clinical, cognitive, and neural phenotypes during acute LLD, which in turn have distinct genotypic correlates.

Specifically, CN individuals will have earlier first onset of depression (EOD) relative to AD, more negative life stress during acute depression compared with AD and PCI, and greater white matter integrity; CN will also be associated with the AA genotype of the COMT val158met polymorphism, which may confer both neuroprotection and higher stress sensitivity. PCI will have more EOD relative to AD, greater frailty, and lower white matter integrity than NC. AD will be associated with later age of depression onset (LOD), greater appetite loss, lower anxiety, smaller hippocampal volume, and greater memory impairment. To test these hypotheses, we propose the following

ELIGIBILITY:
Inclusion Criteria:

For depressed group:

1. Age > 60 years
2. Major depression, single episode or recurrent
3. Ability to read and write English
4. MMSE >25
5. Willingness to participate in the follow-up study for at least two years.

For non-depressed group:

1. Age > 60 years
2. Ability to read and write English
3. MMSE >25
4. Willingness to participate in the follow-up study for at least two years.

Exclusion Criteria:

1. Lifetime alcohol or drug dependence
2. conditions associated with MRI abnormalities such hydrocephalus, benign and cancerous brain tumors, epilepsy, Parkinson's disease, Huntington's chorea, dementia, demyelinating diseases, etc.
3. endocrine disorder other than diabetes mellitus)
4. Any physical or intellectual disability that may affect completion of self rating instruments
5. Established clinical diagnosis of dementia
6. Other primary psychiatric disorders, including panic disorder, social phobia, OCD, non-affective psychosis (including schizo-affective disorder), schizophrenia, bipolar disorder
7. Any metal or pacemaker in the body which precludes MRI.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic Outpatient psychiatry clinic Inpatient psychiatry clinic Self-referral
Sampling Method: Non-Probability Sample
Enrollment: 795 (Actual)
Dates: Start 1995-12; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Depression status (measured by Montgomery Asberg Depression Rating Scale) | Minimum of once per year, up to 21 years
Change in Cognitive impairment (as measuring using cognitive tests including those found in the CERAD battery) | Once per year, up to 21 years
Development of dementia (Determined by Clinical Consensus Conference) | once per year, up to 14 years

SECONDARY OUTCOMES:
Change in Cognition (as measured by tests including those in the CERAD battery) Change in Brain MRI markers (e.g., volume of white matter and gray matter lesions) | once per year, up to 21 years
Change in Impairment in Instrumental or Basic Activities of Daily Living | at least once per year, up to 21 years
Packing density of prefrontal cortex neurons with pyramidal morphology in post-mortem neuroanatomical studies | once post-mortem

CONTACTS AND LOCATIONS:
Overall Officials: Guy G Potter, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Steffens DC, Potter GG, McQuoid DR, MacFall JR, Payne ME, Burke JR, Plassman BL, Welsh-Bohmer KA. Longitudinal magnetic resonance imaging vascular changes, apolipoprotein E genotype, and development of dementia in the neurocognitive outcomes of depression in the elderly study. Am J Geriatr Psychiatry. 2007 Oct;15(10):839-49. doi: 10.1097/JGP.0b013e318048a1a0. Epub 2007 Jul 10. PMID 17623814
- [Result] Steffens DC, Taylor WD, McQuoid DR, Krishnan KR. Short/long heterozygotes at 5HTTLPR and white matter lesions in geriatric depression. Int J Geriatr Psychiatry. 2008 Mar;23(3):244-8. doi: 10.1002/gps.1869. PMID 17702053
- [Result] Potter GG, Blackwell AD, McQuoid DR, Payne ME, Steffens DC, Sahakian BJ, Welsh-Bohmer KA, Krishnan KR. Prefrontal white matter lesions and prefrontal task impersistence in depressed and nondepressed elders. Neuropsychopharmacology. 2007 Oct;32(10):2135-42. doi: 10.1038/sj.npp.1301339. Epub 2007 Feb 14. PMID 17299509
- See also: Longitudinal Geriatric Depression Study — https://clinicaltrials.gov/ct2/show/NCT00570583?term=Duke+Psychiatry&recrs=cd&map_cntry=US&map_state=US%3ANC&rank=2